CLINICAL TRIAL: NCT03910465
Title: Natural History Study of Children and Adults With Chordoma
Brief Title: Children and Adults With Chordoma
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190082; 19-C-0082
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-05-01

CONDITIONS: Chordoma
Keywords: Rare Tumor; Comprehensive Evaluation and Recommendations; Collecting Clinical, Epidemiologic and Biological Data; Natural History
MeSH Terms: conditions — Chordoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Cohort 1: Subjects with confirmed chordoma.

SUMMARY:
Background:

Chordoma is a rare type of bone cancer. It occurs in the skull base or spine. Researchers want to study people with chordoma in different ways. They hope this will help them design better future treatments and supportive care studies for this disease.

Objective:

To learn more about chordoma by looking at its clinical course, how it appears on imagine scans, and how it responds to therapies and treatments.

Eligibility:

People ages 2 and older with chordoma who are enrolled in NCI protocol 19-C-0016

Design:

Participants will be screened with their medical history.

Participants will have a visit to examine their disease. This will include:

* Physical exam
* Neurologic exam
* CT scan and MRI: Participants will lie on a table. The table will slide into a machine. The machine will take pictures of the body.

Participants will have other tests every 6-12 months:

* Smell test
* Surveys to assess their emotional, physical, and behavioral well-being and needs
* Cognitive function tests

Participants or their home doctors will be contacted every 6 12 months. They will be asked to provide information about their disease. This could include test results and imaging evaluations.

Some participants may be asked to come to the clinic for more visits.

DETAILED DESCRIPTION:
Background:

* Chordomas are a rare tumor with an incidence of 325 new cases per year in the United States. Pediatric chordomas are very rare and comprise only 5% of all chordoma cases.
* The standard therapy for localized primary or recurrent chordomas is surgical resection. However, complete surgical resection is often not possible due to the location of the

chordoma.

-For chordomas that cannot be surgically resected, treatment options are limited. Currently,

no standard therapy approach exists for recurrent chordomas. In addition, there are no FDA approved medical therapies for chordoma.

* The natural history of pediatric and adult chordoma is incompletely understood. Patients with chordoma seek expert advice in the management of their care.
* The NCI has basic and clinical expertise and research interest in chordoma. The planned natural history study as part of the NCI POB Rare Tumor Patient Engagement Network (RTPEN) will allow for comprehensive evaluation and recommendations to these patients while longitudinally collecting clinical, epidemiologic and biological data.

Objective:

-To characterize the natural history of chordoma, including clinical presentation and patterns of disease progression.

Eligibility:

* Subjects with radiographically or histologically documented chordoma.
* Age greater than or equal to 2 years old

Design:

-This protocol is a subprotocol to protocol 19-C-0016: Natural History and Biospecimen

Acquisition Study for Children and Adults with Rare Solid Tumors . After enrollment on the master protocol and undergoing evaluations detailed, participants will be enrolled on this subprotocol specific for chordoma.

-Medical histories will be documented, and participants followed throughout the course of their disease, with particular attention to patterns of disease recurrence and progression, response to therapies, duration of responses and patient reported outcomes. Tumor growth rates will also be calculated throughout the course of the disease.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written consent document.
* Subjects with radiographically or histologically documented chordoma
* Age greater than or equal to 2 years old
* Subjects must be enrolled into NCI protocol 19-C-0016: Natural History and Biospecimen Acquisition Study for Children and Adults with Rare Solid Tumors .

EXCLUSION CRITERIA:

-None

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To characterize the natural history of chordoma, including clinical presentation and patterns of disease progression | 10 years
  Natural history of chordoma, including clinical presentation and patterns of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Wedekind Malone, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Derived] Wedekind MF, Widemann BC, Cote G. Chordoma: Current status, problems, and future directions. Curr Probl Cancer. 2021 Aug;45(4):100771. doi: 10.1016/j.currproblcancer.2021.100771. Epub 2021 Jul 1. PMID 34266694
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0082.html